CLINICAL TRIAL: NCT00444886
Title: Treatment of Thoracic Outlet Syndrome With Botulinum Toxin Injection: A Double-Blind, Randomized Controlled Trial
Brief Title: Treatment of Thoracic Outlet Syndrome (TOS) With Botox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Allergan (Industry)
Responsible Party: Heather Finlayson, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H06-03355; Data not known
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Thoracic Outlet Syndrome (TOS); Botulinum Toxin; Botox; Pain
MeSH Terms: conditions — Thoracic Outlet Syndrome; Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): To assess the effect of BOTOX injection to the scalene muscles on the severity of pain from TOS.
  Interventions: Drug: Botulinum Toxin Type A injection (BOTOX)
- 2 (Active Comparator): To assess the effect of BOTOX injection on numbness and tingling and quality of life.
  Interventions: Drug: Botulinum Toxin Type A injection (BOTOX)

INTERVENTIONS:
Drug: Botulinum Toxin Type A injection (BOTOX) — Each subject will receive an injection under EMG guidance into the anterior and middle scalene muscles of either 75 units of BTX-A (experimental group), or normal saline (control group). Both groups will be provided with a stretching and strengthening exercise program.
  Arms: 1
Drug: Botulinum Toxin Type A injection (BOTOX) — Each subject will receive an injection under EMG guidance into the anterior and middle scalene muscles of either 75 units of BTX-A (experimental group), or normal saline (control group). Both groups will be provided with a stretching and strengthening exercise program.
  Arms: 2

SUMMARY:
The purpose of this study is:

1. To assess the effect of BOTOX injection to the scalene muscles on the severity of pain from TOS.
2. To assess the effect of BOTOX injection on numbness and tingling and quality of life.

DETAILED DESCRIPTION:
Background:

Thoracic Outlet Syndrome (TOS) is a symptom complex consisting of pain, paresthesias and often functional impairment caused by compression of the neurovascular supply to the upper limb. Impingement may occur at the interscalene triangle, and both anesthetic blockade and chemodenervation of the scalene muscles have been shown to temporarily improve symptoms of TOS in non-randomized controlled trials.

Objective:

To assess the effect of Botulinum Toxin Type A (BTX-A) injections into the scalene muscles on pain, paresthesias and function in subjects with TOS.

Hypothesis:

BTX-A injected into the anterior and middle scalene muscles will reduce the irritation on the neurovascular structures at the interscalene triangle in subjects with TOS. This will lead to reductions in pain and paresthesias, and improvements in function when compared with injection of placebo.

Intervention:

Each subject will receive an injection under EMG guidance into the anterior and middle scalene muscles of either 75 units of BTX-A (experimental group), or normal saline (control group). Both groups will be provided with a stretching and strengthening exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 19 years
* Medically stable
* Able to give informed consent
* Meets criteria for clinical diagnosis of TOS
* Symptoms of TOS present for at least six months
* Have had EMG studies and a CT or MRI scan of the cervical spine

Exclusion Criteria:

* Prior treatment with BTX-A
* Allergy to BTX-A
* History of botulinum toxicity
* Prior scalenectomy
* Surgery for TOS planned within six months
* Use of blood thinners, i.e., warfarin; unfractionated or low molecular weight heparin
* History of Myasthenia Gravis, Eaton-Lambert Syndrome or Shy-Drager Syndrome
* Unable to complete follow-up assessments at 6 weeks, 3 months and 6 months
* Any abnormalities on EMG, CT or MRI studies suggesting an alternate diagnosis
* Pregnancy or planned pregnancy within six months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pain as measured on Visual Analog Scale (VAS) at 6 weeks, 3 months and 6 months post-intervention | 6 monhts

SECONDARY OUTCOMES:
Paresthesias as measured on VAS | 6 months
Function as measured with Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, SF-36, number of days lost from work | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Travlos, MD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada